## Physical ACtivity Enhancement Scheme (PACES) in hemodialysis patients: a cross-sectional investigation

Ethics Committee Approval (No 20211575)

Investgator Mei Huang

Version 1 Edited on 1 September 2021

## **Informed Consent Forms**

Dear participant:

Hello!

This study is a key research and development project of Shaanxi Province. The purpose of the study is to understand your physical activity status and explore relevant influencing factors, so as to provide a basis for the development of Physical ACtivity Enhancement Scheme (PACES) for you in the next stage, so that we can solve your doubts about PA and establish the right perception of PA so that you can PACE to improve PA.

It will take you about 10 minutes to fill in these questionnaires. Please fill it carefully according to your actual situation.

The information you provided is only used for this study, we will not disclose to any institutions or individuals, please rest assured!

Thank you very much for your participation!

| Research | er's signatu | re: | |
|-----------|--------------|-------|-----|
| Patient s | signature: | | |
| Date: | year | month | day |